CLINICAL TRIAL: NCT06559371
Title: 68Ga FAPI PET/CT Evaluation of Axillary Lymph Node Status After Neoadjuvant Therapy in Patients With Clinical Axillary Lymph Node Positive Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Kunwei Shen (Other)
Responsible Party: Sponsor-Investigator, Kunwei Shen, Professor, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Other Study IDs: RJBC-2403
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-08

CONDITIONS: BREAST CANCER; PET/CT
Keywords: BREAST CANCER; PET/CT
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 68Ga-FAPI PET/CT: 68Ga-FAPI PET/CT

SUMMARY:
The goal of this observational study is to learn whether 68Ga-FAPI PET/CT may be used as a new effective methods for evaluating axillary lymph node efficacy after neoadjuvant treatment for breast cancer. The main question it aims to answer is:

Could 68Ga-FAPI PET/CT effectively evaluate axillary lymph node after neoadjuvant treatment for breast cancer? Participants will have a 68Ga-FAPI PET/CT test between last neoadjuvant therapy and surgery.

DETAILED DESCRIPTION:
Previous studies have shown that compared with conventional 18F-FDG PET/CT, 68Ga-FAPI PET/CT has the characteristics of not being affected by blood glucose, good tumor specificity, and high tumor-to-background ratio, and studies have shown that 68Ga- FAPI PET/CT can detect parts of breast cancer primary lesions and lymph node metastases with low 18F-FDG uptake, thereby increasing the lesion detection rate and improving the sensitivity of imaging examinations. Therefore, 68Ga-FAPI PET/CT may be used as a new effective methods for evaluating axillary lymph node efficacy after neoadjuvant treatment for breast cancer. Therefore, we plan to conduct this study to explore the ability of 68Ga-FAPI PET/CT to detect residual disease in axillary lymph nodes in patients with clinically positive axillary node (cN+) breast cancer after neoadjuvant treatment. By this way, we may explore an accurate and non-invasive assessment of axillary lymph node status after neoadjuvant therapy in breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 and above
* ECOG score 0-2 points
* Pathological confirmation of malignant breast tumor
* Clinical axillary lymph node positivity (cN+)
* Completed at least 3 courses of neoadjuvant therapy and subjected to undergo surgical treatment
* Informed consent form signed

Exclusion Criteria:

* Distant metastasis
* Unable to complete the proposed neoadjuvant therapy plan
* Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Female patients aged 18 and above
  * ECOG score 0-2 points
  * Pathological confirmation of malignant breast tumor
  * Clinical axillary lymph node positivity (cN+)
  * Completed at least 3 courses of neoadjuvant therapy and subjected to undergo surgical treatment
  * Informed consent form signed
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of 68Ga FAPI PET/CT in predicting residual axillary lymph node lesions after neoadjuvant therapy | up to the end of surgery
  Sensitivity and specificity of 68Ga FAPI PET/CT

SECONDARY OUTCOMES:
Sensitivity and specificity of 68Ga FAPI PET/CT in predicting pathological complete response (Breast pCR) of breast lesions in neoadjuvant therapy | up to the end of surgery
  Sensitivity and specificity of 68Ga FAPI PET/CT in predicting pathological complete response (Breast pCR) of breast lesions in neoadjuvant therapy
Sensitivity and specificity of 68Ga FAPI PET/CT in predicting objective response rate (ORR) of neoadjuvant therapy | up to the end of surgery
  Sensitivity and specificity of 68Ga FAPI PET/CT in predicting objective response rate (ORR) of neoadjuvant therapy
68Ga FAPI PET/CT in predicting invasive disease free survival after neoadjuvant therapy | From enrollment to the end of treatment at 3 years
  68Ga FAPI PET/CT in predicting invasive disease free survival after neoadjuvant therapy
68Ga FAPI PET/CT in predicting overall survival after neoadjuvant therapy | From enrollment to the end of treatment at 3 years
  68Ga FAPI PET/CT in predicting overall survival after neoadjuvant therapy

CONTACTS AND LOCATIONS:
Overall Officials: Xiaosong Chen, Principal Investigator — Shanghai Jiao Tong University, School of Medicine, Affiliated Ruijin Hospital
Locations (1):
- Shanghai Jiao Tong University School of Medicine, Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No